CLINICAL TRIAL: NCT01313884
Title: A Phase II Pilot Study of Cyclophosphamide, Doxorubicin, Vincristine Alternating With Irinotecan and Temozolomide in Patients With Newly Diagnosed Metastatic Ewing's Sarcoma
Brief Title: Cyclophosphamide, Doxorubicin, Vincristine w/ Irinotecan and Temozolomide in Ewings Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not reach primary objective; study did not accrue enough patients.
Sponsor: Stanford University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Kristen Ganjoo, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20323; SU-03082011-7559 (Other: Stanford University); SARCOMA0007 (Other: OnCore)
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2016-12

CONDITIONS: Bone Cancer; Ewing's Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Sarcoma, Ewing | interventions — Irinotecan; Vincristine; Temozolomide; Doxorubicin; Cyclophosphamide; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Therapy (Experimental): Regimen A alternating with Regimen B every 21 days
  Regimen A:
  * Cytoxan 1200mg/m2
  * Doxorubicin, starting dose 75 mg/m2 to a maximum of 450mg/m2
  * Vincristine, starting dose 2 mg/m2 to a maximum of 2 mg
  * Pegfilgrastim, 6 mg subcutaneous within 24 to 48 hours after each cycle
  Regimen B:
  * Irinotecan 50 mg/m2/day x 5 days
  * Temozolomide 100 mg/m2/day x 5 days followed by 2 weeks treatment-free
  Interventions: Drug: Irinotecan; Drug: Vincristine; Drug: Temozolomide; Drug: Doxorubicin; Drug: Cytoxan; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Irinotecan — 50 mg/m2/day x 5 days
  Other Names: Camptosar; Campto
Drug: Vincristine — 2 mg/m2 to a maximum of 2 mg
  Other Names: Oncovin; leurocristine
Drug: Temozolomide — 100 mg/m2/day x 5 days followed by 2 weeks treatment-free
  Other Names: Temodar; Temodal
Drug: Doxorubicin — Starting dose 75 mg/m2 to a maximum of 450mg/m2
  Other Names: Adriamycin; hydroxydaunorubicin
Drug: Cytoxan — 1200 mg/m2
  Other Names: Cyclophosphamide; Endoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Pegfilgrastim — 6 mg subcutaneous within 24 to 48 hours after each Regimen A cycle
  Other Names: Neulasta

SUMMARY:
The outcome of patients with metastatic Ewings Sarcoma is poor with current standard of care chemotherapy, with less than 30% survival. Based on recent encouraging pediatric literature we have designed this trial to improve the outcome of patients with metastatic Ewings sarcoma using Irinotecan and Temozolomide in addition to standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic Ewing's sarcoma.
* Patients must have measurable disease defined as lesions that can be measured by medical imaging techniques such as CT or MRI. Ascites, pleural fluid, bone marrow disease, lesions seen on scan will not be considered measurable.
* Patients must have metastatic disease.
* Age 13 years or older
* Life expectancy of at least 3 months.
* ECOG performance status of <= 3.
* Normal hepatic function (Direct bilirubin <1.5mg/dl, SGOT or SGPT <3x upper limit of normal).
* Left Ventricular Ejection fraction of at least 50%.
* Adequate renal function: Creatinine clearance >= 50 ml/min or Serum creatinine < 1.5 x ULN for age.
* Adequate bone marrow reserve (defined as an absolute peripheral granulocyte count of >=1500/mm3, platelet count of >=75,000/mm3); unless bone marrow infiltrated with metastatic Ewing's sarcoma; ANC >= 500 and Platelet >= 50,000 mm3.
* Ability to understand and willing to sign a written informed consent document.
* Patients of childbearing potential must agree to use an effective method of contraception.

Exclusion Criteria:

* No prior chemotherapy for Ewing's sarcoma; No prior doxorubicin, temozolomide or irinotecan.
* Known hypersensitivity to any of the components of the protocol drugs.
* Clinically significant unrelated systemic illness (such as serious infections requiring active systemic intravenous antibiotic therapy; cardiovascular disease [congestive heart failure, recent myocardial infarction, unstable angina, inadequately controlled hypertension].
* No prior history of chronic diarrhea, bowel obstruction, Crohn's disease or ulcerative colitis.
* Pregnant or nursing woman are not included in the study.
* HIV-positive patients will be excluded from the study due to risk of infection or other serious side effects.
* Other medical, psychiatric or social condition incompatible with study treatment.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N. Ganjoo, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy: Regimen A alternate with Regimen B every 21 days
  Regimen A:
  Cytoxan=1200mg/m2 Doxorubicin=75mg/m2 (Maxiumum allowed dose 450mg/m2) Vincristine=2mg/m2 (capped at 2mg total dose)
  Regimen B:
  Irinotecan=50 mg/m2/day x 5 days Temozolomide=100 mg/m2/day x 5 days followed by two weeks of treatment-free period.
  Irinotecan: 50 mg/m2/day x 5 days
  Vincristine: 2 mg/m2 (capped at 2mg total do)
  Temozolomide: 100 mg/m2/day x 5 days
  Doxorubicin: 75 mg/m2
  Cytoxan: 1200 mg/m2
  Pegfilgrastim: 6 mg
  Mesna: 240 mg/m2 in 50 ml NS
Period: Overall Study
Arm/Group | Combination Therapy
Started | 3
Completed | 2
Not Completed | 1
Not completed — Per insurance pvdr, pt can't be on cl tr | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Partial and Complete Response)
Description: Response was evaluated every 12 weeks during treatment. Subjects who discontinue treatment for reasons other than disease progression or initiation of new anticancer therapy (excluding radiation therapy and surgery) response evaluated every 6 months following the last dose of study drug. Scans should be obtained every 6 months for up to 2 years (24 months) or until progression of disease or initiation of new anticancer therapy.
  Complete response (CR) Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as a reference the baseline sum diameters.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 2
Participants
  Complete Response | 0
  Partial Response | 2

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The intended outcome is a measure of whether participants are alive without disease progression 2 years (24 months) after treatment.
Time Frame: 24 months
Population: All study participants were lost to follow-up after completion of active treatment and collection of response rate, ie, within 2 years of the treatment conclusion but before documented progression. No data.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All adverse events (related and unrelated) occurring during the study (from the time the patient receives the first dose of study drug) and up to 30 days after the last dose of study medication were reported.
Description: Patients were asked about adverse events at every clinic visit.
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=3)
Intermittent headache G1 (General disorders) | 1 (1)
Decreased energy G1 (Gastrointestinal disorders) | 1 (1)
Fatigue G1 (Gastrointestinal disorders) | 1 (1)
Insomnia G1 (General disorders) | 1 (1)
Insomnia G2 (General disorders) | 1 (1)
Fever G1 (General disorders) | 1 (1)
Hiccups G1 (General disorders) | 1 (1)
Throat pain G2 (Gastrointestinal disorders) | 1 (1)
Nausea G1 (Gastrointestinal disorders) | 1 (1)
Nausea, intermittent G1 (Gastrointestinal disorders) | 1 (1)
Nausea, intermittent G2 (Gastrointestinal disorders) | 1 (1)
Mucositis oral G1 (Gastrointestinal disorders) | 2 (2)
Oral lesions G1 (Gastrointestinal disorders) | 1 (1)
oral candidiasis G1 (Gastrointestinal disorders) | 1 (1)
Sore throat G1 (Gastrointestinal disorders) | 1 (1)
Pain with swallowing G1 (Gastrointestinal disorders) | 1 (1)
Worsening acid reflux G1 (Gastrointestinal disorders) | 1 (1)
Diarrhea G1 (Gastrointestinal disorders) | 2 (3)
Abdominal cramping G1 (Gastrointestinal disorders) | 1 (1)
Abdominal pain G1 (Gastrointestinal disorders) | 1 (1)
Intermittent diarrhea G1 (Gastrointestinal disorders) | 1 (1)
Vomiting G1 (Gastrointestinal disorders) | 1 (1)
Vomiting intermittent G1 (Gastrointestinal disorders) | 1 (1)
Constipation G1 (Gastrointestinal disorders) | 1 (1)
Nausea and vomiting G1 (Gastrointestinal disorders) | 1 (1)
Anemia G2 (Blood and lymphatic system disorders) | 1 (2)
Worsened anemia G2 (Blood and lymphatic system disorders) | 1 (1)
Anemia G3 (Blood and lymphatic system disorders) | 1 (1)
Decreased neutrophils G4 (Blood and lymphatic system disorders) | 1 (1)
Infection-staph epidermis bacteremia (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased G1 (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia G1 (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia intermittent G1 (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia intermittent G1 (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased G2 (Blood and lymphatic system disorders) | 1 (2)
Platelet count decreased G4 (Blood and lymphatic system disorders) | 1 (1)
Intermittent hypoglycemia G1 (Metabolism and nutrition disorders) | 1 (1)
White blood cells decreased G2 (Blood and lymphatic system disorders) | 1 (1)
White blood cells decreased G4 (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia G1 (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia G1 (Metabolism and nutrition disorders) | 1 (1)
Hip pain L G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain sacrum (tailbone) G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain left leg G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-lowe leg, back G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain generalized 2-3 days post neulasta G1 (General disorders) | 1 (1)
Tingling at left toes G1 (Nervous system disorders) | 1 (1)
Numbness on left shin G1 (Nervous system disorders) | 1 (1)
Cough G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Onychomycosis G2 (Skin and subcutaneous tissue disorders) | 1 (1)
Hip abscess G3 (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema L hip G2 (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema groin crease G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema left leg G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Edema left leg pitting 2+, G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperpigmentation left knee G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Disc edema R eye G1 (Eye disorders) | 1 (1)
Nasal congestion G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study did not reach primary objective; study didn't accrue enough patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes